CLINICAL TRIAL: NCT05211713
Title: Opp: The Development and Evaluation of a Mental Health App for Adolescents
Brief Title: Opp - a Universal Mental Health Promoting Mobile Application for Adolescents
Acronym: Opp
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: The Dam Foundation (Other); Norwegian Council for Mental Health (Other); Norwegian Directorate of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 279207
Record Dates: First submitted 2021-12-15; First posted 2022-01-27 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Mental Health Wellness 1
Keywords: Mental health promotion; Coping; Adolescents; Mobile application

STUDY DESIGN:
Intervention Model Description: Intervention and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group receiving Opp (Experimental): The effectiveness study will be conducted as a randomized controlled trial with an intervention group and a waiting-list control group. Data will be collected at baseline (T1, pre intervention) and after about six weeks of intervention (T2, post intervention).
  Interventions: Device: Opp
- Control group (No Intervention): The waiting list control group will receive the intervention after study completion.

INTERVENTIONS:
Device: Opp — Opp is a universal mental health promoting mobile application for adolescents aged 13-25 years.
  Arms: Intervention group receiving Opp

SUMMARY:
The aim of the project is firstly, to develop an app-based mental health intervention for adolescents. Secondly, to evaluate the effect of this app. The overarching goal is to offer a low-threshold intervention, called Opp, that is easily accessible and free to use for all adolescents in Norway.

DETAILED DESCRIPTION:
The intervention "Opp" will be delivered through a mobile application. The overall goals of Opp are to 1) increase well-being and mental well-being, 2) increase knowledge about mental health, 3) increase coping skills to deal with stress, 4) increase help-seeking behavior, 5) increase self-esteem, 6) increase sleep quality and 7) reduce mental health problems.

To evaluate the mobile application two studies will be conducted: A user survey and an effectiveness study with a follow-up examination after about six weeks. The effectiveness study will be conducted as a randomized controlled trial with an intervention group and a waiting-list control group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents under 16 years whose guardians have given consent

Exclusion Criteria:

* severe developmental or cognitive challenges

Ages: 13 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in WHO-5 (WHO-Five Well-being Index) | Change from baseline to six weeks after intervention.
  WHO-5 (WHO, 1998): A five item self-report questionnaire assessing well-being on a six point scale.
Change in SDQ (Strengths and Difficulties Questionnaire) | Change from baseline to six weeks after intervention.
  SDQ (Goodman, 1997): A 25 item self-report assessing mental health and psychosocial functioning in 11-17 years old adolescents on a three point scale.

SECONDARY OUTCOMES:
General Self-efficacy scale (GSE) | Change from baseline to six weeks after intervention.
  Resilience will be measured with the Norwegian version of the GSE (Røysamb, 1997; Schwarzer et al., 1995) which consists of 10 questions measured on a four-point scale.
Help-seeking behavior | Change from baseline to six weeks after intervention.
  Two self-report items measuring if they sought help and who they sought help from.
Self-liking and Competence Scale | Change from baseline to six weeks after intervention.
  Self-liking and Competence Scale (Silvera, Neilands, & Perry, 2001; Tafarodi & Swann, 2001): A 20 item self-report assessing self-liking and self-competence.
Sleeping quality | Change from baseline to six weeks after intervention.
  Sleeping quality will be measured with six questions from the Bergen Child Study (Hysing, Harvey, Stormark, Pallesen, & Sivertsen, 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Henriette Kyrrestad, PhD, Principal Investigator — UiT The Arctic University of Norway
Locations (1):
- UiT The Arctic University of Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaiser S, Rye M, Jakobsen R, Martinussen M, Hogsdal H, Kyrrestad H. A Universal Mental Health-Promoting Mobile App for Adolescents: Protocol for a Cluster Randomized Controlled Trial. JMIR Res Protoc. 2023 Jan 11;12:e42119. doi: 10.2196/42119. PMID 36630167
- See also: Homepage — http://uit.no/forskning/opp